CLINICAL TRIAL: NCT02302001
Title: Breast Augmentation Using Novel Method of Jet Hydro Dissection Effects on Postoperative Pain
Brief Title: Effects of Jet Hydro Dissection in Breast Augmentation Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristocrat Plastic Surgery and MedAesthetics (Other)
Collaborators: Erbe-med (Unknown); Tiger Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fwa00022532
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Breast Augmentation
Keywords: Breast augmentation; Breast implants; Silicone implants; Breast surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Primary Breast Augmentation (Experimental)
  Interventions: Device: Silicone Implant

INTERVENTIONS:
Device: Silicone Implant

SUMMARY:
ERBEjet Breast augmentation is a novel method of dissection of the subpectoral pocket. Study is designed to differentiate parameters of pain between randomized laterality using no touch technique. THIS IS NOT A FREE STUDY. Patients are required to pay the initial cost of surgery but will receive a refund of a partial payment. Patients must undergo evaluation at consultation and surgical quote is provided.

DETAILED DESCRIPTION:
Breast augmentation in the subpectoral position has classically been associated with postoperative pain and discomfort within the first two weeks after the operation. Minimizing this pain and discomfort and ability to return to normal function soon after the operation has been the goal of numerous interventions. Minimal injury no touch dissection techniques have proven results regarding morbidity. ERBEjet is a novel dissection using a jet of local anesthetic infused saline fluid with a built in coagulation function used for dissection of soft tissues. The study is designed to randomly perform ERBEjet Breast augmentation operation unilaterally on breast augmentation and mastopexy augmentation patients undergoing traditional sub pectoral dissection technique on the contralateral side. Patient's record pain scores at regular intervals in the postoperative period. Physical examination performed by blinded practitioners assess discomfort and tenderness scores within the two weeks after the operation.

ELIGIBILITY:
Inclusion Criteria:

* silicone breast implants candidate

Exclusion Criteria:

* history of breast cancer
* inability to conform to post operative questionnaire and recovery follow up

Ages: 22 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Decreased postoperative pain and recovery after breast augmentation | Two weeks

SECONDARY OUTCOMES:
Decreased risk of capsular contracture | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Tehrani, M.D., Principal Investigator — Aristocrat Plastic Surgery
Locations (2):
- United States (2):
  - Aristocrat Plastic Surgery & MedAesthetics, Great Neck, New York
  - Aristocrat Plastic Surgery, New York, New York